CLINICAL TRIAL: NCT05288803
Title: Improving Rehabilitation for Veterans After Total Knee Arthroplasty Using Individualized Recovery Trajectories
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F3770-R; I01RX003770 (NIH)
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Arthroplasty
Keywords: total knee arthroplasty; patient-centered care; precision medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control cohort: The investigators will collect outcomes for 100 Veterans treated with usual care rehabilitation after total knee arthroplasty. Data will be collected at all participating clinical locations. Data collection for these Veterans will precede data collection for the intervention cohort.
- Intervention cohort: The investigators will implement the clinical decision support tool in all participating clinic locations. We will collect outcomes for 100 Veterans treated in rehabilitation with use of the clinical decision support tool. Data collection for these Veterans will occur after data collection is complete for the Control cohort.
  Interventions: Other: Clinical decision support tool (CDS tool)

INTERVENTIONS:
Other: Clinical decision support tool (CDS tool) — The investigators will integrate the CDS tool into clinical practice at each participating clinic after data collection for the Control cohort is complete. All physical therapists at the participating clinic locations will use the CDS tool to inform rehabilitation decision making for Veterans with total knee arthroplasty. The CDS tool will provide personalized information regarding each Veterans' recovery in addition to personalized visit utilization guidelines. Clinicians will use the CDS tool with Veterans at their initial postoperative visits and every 2weeks throughout their course of care thereafter.
  Other Names: Knee Recovery Tool
  Groups: Intervention cohort

SUMMARY:
This study will examine the impact of a new clinical decision support tool for rehabilitation after total knee arthroplasty (TKA). Typically, TKA rehabilitation is generic with most patients receiving the same dosage and contents of rehabilitation despite notable diversity among patients who undergo TKA. The investigators clinical support decision tool is designed to help physical therapists tailor rehabilitation treatments and dosages to the individual needs, goals, and preferences of Veterans recovering from TKA. This study has the potential to improve Veterans' functional recovery after TKA, while simultaneously reducing the average number of physical therapy visits Veterans attend after surgery by tailoring rehabilitation dosage based upon need. This will ensure the Veterans Health Administration (VHA) has the resources and capacity to provide adequate rehabilitation to every Veteran seeking TKA in the VHA system. Additionally, if successful, this clinical decision support tool could be used to improve outcomes and access for additional patient populations in the future.

DETAILED DESCRIPTION:
Rehabilitation after total knee arthroplasty (TKA) is typically generic and inefficient; most patients receive the same contents and dosage of rehabilitation regardless of the patients individual needs, preferences, or expectations. This generic treatment paradigm will be unsustainable in the Veterans Health Administration (VHA) as the demand for TKA surgery and postoperative care increase exponentially in the near future. Without new strategies to improve the efficiency of TKA rehabilitation, organizations like the VHA will struggle to meet and pay for this surging demand, and Veterans may be denied timely access to the postoperative care they need for optimal recovery. The investigators have developed an innovative new clinical decision support (CDS) tool to optimize efficiency in TKA rehabilitation. Using the actual recovery data of similar historical patients, the tool can predict the recovery trajectory for new patients after TKA. This allows clinicians to (1) allocate rehabilitation resources based upon individual need, (2) identify Veterans at risk for suboptimal outcomes early after surgery, (3) tailor treatment strategies to Veterans' unique goals and clinical presentation, and (4) monitor Veterans' recovery relative to expected throughout postoperative rehabilitation. In this project, the investigators propose to expand the CDS tool's capabilities by establishing utilization guidelines based upon individual Veteran's predicted recovery (Aim 1). These guidelines will be established by expert consensus in a three round Delphi process. Subsequently, the investigators will test the CDS tool's impact on Veteran's functional recovery and rehabilitation utilization in four VHA outpatient physical therapy clinics using a pre-post design (Aim 2). The investigators will compare patient-reported function (Lower Extremity Functional Scale) and physical therapy visit utilization between cohorts of Veterans treated with and without the CDS tool. Additionally, the investigators will gather data from participating VHA clinicians and Veterans regarding the translation of the investigators tool into clinical practice to assess its readiness for dissemination throughout the VHA (Aim 3). This will include qualitative data from participant focus groups and quantitative process data regarding the tool's utilization. Ultimately, the investigators expect this study will serve as a template for expanding the investigators tool's capabilities into numerous VHA populations in rehabilitation and beyond.

ELIGIBILITY:
Inclusion Criteria:

-Veterans who have undergone total knee arthroplasty who present for outpatient rehabilitation treatment at the participating clinics within three weeks of surgery.

Exclusion Criteria:

* postoperative rehabilitation treatment received in the home health or skilled nursing
* age < 40 or >90

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with total knee replacement who seek postoperative outpatient physical therapy treatment at the participating clinics.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome - Joint Replacement (KOOS, JR) | Change in KOOS Jr from preop (baseline) to postop (90 days after TKA surgery)
  The KOOS-JR is a patient-reported measure of physical function developed specifically for patients with total knee arthroplasty. It can be completed quickly (only 7 items) and has established validity, reliability, and responsiveness. KOOS JR will also be assessed at 30, 60, and 180 days after TKA surgery. We will use the interval scoring method for the KOOS JR which ranges from 0 (total knee disability) to 100 (perfect knee health)
Outpatient Physical Therapy Visit Utilization | Postoperative day 90
  The total outpatient physical therapy visits used in the first 90 postoperative days by each Veteran participant will be extracted from the electronic health record after the Veteran is formally discharged from outpatient rehabilitation. Any visits that occur prior to a Veteran's surgery or in the hospital setting will not count toward the total visit number. We chose postoperative day 90 as our primary endpoint because it corresponds with the average discharge timeframe for outpatient rehabilitation after total knee arthroplasty. Visit utilization will also be assed at at 30, 60, and 180 days after TKA surgery.

SECONDARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | Change in LEFS from preop (baseline) to postop (90 days after TKA surgery).
  The LEFS is a generic scale of lower extremity physical function that has established validity, reliability, and sensitivity to change for patients with total knee arthroplasty. LEFS will also be assessed at 30, 60, and 180 days after TKA surgery. The LEFS scale ranges from 0 (lowest function) to 80 (highest function).
Timed Up and Go (TUG) | Change in TUG from preop (baseline) to postop (90 days after TKA surgery)
  The TUG is a basic measure of mobility and balance which consists of rising from a seated position, walking three meters, and pivoting and returning to the original seated position. The TUG is responsive to change with adequate reliability in the acute recovery period after total knee arthroplasty. TUG will also be assessed at 30 and 60 days after TKA surgery.
Knee range of motion (ROM) | Change in knee ROM from preop (baseline) to postop (90 days after TKA surgery)
  Knee ROM will be measured manually by goniometry which is a valid and reliable technique for measuring knee mobility. Recovery of knee ROM after TKA is necessary for many functional activities and is emphasized in rehabilitation after total knee arthroplasty. ROM will also be assessed at 30 and 60 days after TKA surgery.
Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale | Change in WOMAC pain subscale from preop (baseline) to postop (90 days after TKA surgery)
  The WOMAC pain subscale is a valid, reliable, and responsive measure of patient-reported pain for individuals with osteoarthritis of the knee. WOMAC pain subscale will also be assessed at 30 and 60 days after TKA surgery. The WOMAC pain subscale scores range from 0 (lowest pain) to 20 (highest pain).

OTHER OUTCOMES:
Veterans Rand 12-item Health Survey (VR-12) | Collected at preop (baseline) and 90 days after TKA surgery
  The VR-12 mental component summary score will be used to capture emotional/psychosocial variables which could impact Veteran recovery and/or healthcare utilization after total knee arthroplasty. The VR-12 mental component summary score will be included as a potential confounder in our Aim 2 analysis plan. VR-12 will also be assessed at 30 and 60 days after TKA surgery. The VR-12 includes both a Mental Component Score (MCS) and Physical Component Score (PCS). Both scores can be reported as z-scores for the population average in the United States. The population average for both scores is 50, and each 10-point increment above or below 50 corresponds to 1 standard deviation away from the population average.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The research team guarantees that all data collected as part of this project will be released in accordance with standard data sharing policies and procedures to validate research findings if requested. All data released will be de-identified, with no information that could be linked to any study participants (patients and clinicians), or participating study practices to ensure the confidentiality of all participants and practices. If necessary, a data use agreement will be established.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after the main study results are published.
Access Criteria: Data will be available after the main study results are published for up to 5 years.